CLINICAL TRIAL: NCT02046798
Title: An Open Label Study to Evaluate the Pharmacokinetics of ASP3652 After a Single Oral Dose of 14C-labeled ASP3652 in Healthy Caucasian Male Subjects
Brief Title: A Study to Assess the Pharmacokinetics, Metabolism and Excretion Routes of ASP3652 in Man, After Administration of 14C Radio Labeled ASP3652
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 3652-CL-0003; 2011-004526-10 (EudraCT Number)
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Healthy Subjects; Pharmacokinetics of ASP3652
Keywords: Pharmacokinetics; ASP3652; 14C radio-labeled; Phase 1
MeSH Terms: interventions — ASP3652

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 14C labeled ASP3652 (Experimental)
  Interventions: Drug: ASP3652

INTERVENTIONS:
Drug: ASP3652 — oral

SUMMARY:
This study measures how much of the trial drug enters the body and how long it takes for the body to remove it via the feces and urine. In addition, the different breakdown products after a single oral dose of radio-active ASP3652 will be identified.

DETAILED DESCRIPTION:
This is an open-label, one-period, single-dose study with 14C labeled ASP3652.

Screening takes place between Day 22 to Day 2, and subjects are admitted to the clinic on Day -1.

On the morning of Day 1, each subject receives a single oral dose of 14C-labeled ASP3652. Blood, urine and feces samples for analysis of 14C radioactivity are collected until at least 120 h after dosing. Blood samples for the analysis of ASP3652 and metabolites are collected until 120 h after dosing.

The subjects remain in the clinic until Day 6 (or up to Day 13 in case discharge criteria are not met on Day 6) and return for an End of Study Visit (ESV) 7 to 14 days after (early) discharge.

ELIGIBILITY:
Inclusion Criteria:

* Subject is white and of Caucasian origin.
* Regular defecation pattern (minimum once per day).
* Subject must agree to use a condom during sexual intercourse until 3 months after dosing. In addition to using a condom, subjects must agree to practice an adequate contraceptive method with female sexual partners to prevent pregnancy.

Exclusion Criteria:

* Known or suspected hypersensitivity to ASP3652 or any components of the formulation used.
* Donation of blood or blood products within 3 months prior to admission to the Clinical Unit.
* Exposure to radiation for diagnostic reasons (except dental X-rays and plain X-rays of thorax and bony skeleton (excluding spinal column)), during work or during participation in a clinical study in the previous year.

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Total radioactivity in plasma | Days 1 to 6 and up to Day 9
  area under the plasma concentration (AUC) - time curve from time zero to infinity (AUCinf), area under the plasma concentration - time curve from time zero to time of last measurable concentration (AUClast), maximum concentration (Cmax), time to attain Cmax (tmax), apparent terminal elimination half-life (t½)
Total radioactivity in whole blood | Days 1 to 6 and up to Day 9
  area under the plasma concentration (AUC) - time curve from time zero to infinity (AUCinf), area under the plasma concentration - time curve from time zero to time of last measurable concentration (AUClast), maximum concentration (Cmax), time to attain Cmax (tmax), apparent terminal elimination half-life (t½)
Radioactivity ratio of plasma / blood | Days 1 to 6 and up to Day 9
  ratio concentrations per time point and AUC
Radioactivity excretion in urine | Urine: Days 1-6 and up to Day 25
  excretion rate and cumulative excretion
Radioactivity excretion in feces | Days 1-6 and up to Day 25
  excretion rate and cumulative excretion
Radioactivity excretion in urine and feces | Urine: Days 1-6 and up to Day 25
  excretion rate and cumulative excretion
ASP3652 in plasma | Days 1 to 6 and up to Day 9
  AUCinf, AUClast, Cmax, tmax, t1/2, apparent clearance after oral administration at steady state (CL/F), volume of terminal phase distribution at steady state (Vz/F)
ASP3652 in urine | Days 1-6 and up to Day 25
  cumulative amount of unchanged drug excreted into the urine from time zero to infinity after single dose (Aeinf), cumulative amount of unchanged drug excreted into the urine from time zero to time of last measurable concentration (Aelast), renal clearance of the drug from plasma (CLR), percentage of unchanged drug excreted into the urine from time zero to infinity after single dose % of dose excreted (Aeinf%), percentage of unchanged drug excreted into the urine from time zero to time of last measurable concentration (Aelast%)
Ratio ASP3652 to 14C-radioactivity for AUCinf | Days 1 to 6 and up to Day 9
  area under the plasma concentration (AUC) - time curve from time zero to infinity (AUCinf)

SECONDARY OUTCOMES:
Safety and tolerability after a single dose | Screening (Day 22 to Day 2) to End of Study Visit (7 to 14 days after (early) discharge)
  Vital signs, 12-lead ECG, safety laboratory tests, physical examination, occurrence of Adverse Events (AE)

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- Covance Clinical Research Unit (CRU) Ltd., Leeds, United Kingdom